CLINICAL TRIAL: NCT06130124
Title: S-amlodipine in Essential HypertensIon and Assessment of Blood Pressure Targets Achievement According to 2022 KSH(Korean Society of Hypertension) Guidelines (SHIFT)
Brief Title: S-amlodipine in Essential HypertensIon and Assessment of Blood Pressure Targets Achievement
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hanlim Pharm. Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: HL-LDN-403
Record Dates: First submitted 2023-11-08; First posted 2023-11-14 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-07

CONDITIONS: Essential Hypertension
MeSH Terms: conditions — Essential Hypertension

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Evaluate the ratio(%) of patients whose blood pressure measured at 6 months from the baseline was confirmed to be within the target blood pressure range according to the 2022 hypertension treatment guidelines for essential hypertension patients who received the study drug.

DETAILED DESCRIPTION:
Primary purpose:

Evaluate the ratio(%) of patients whose blood pressure measured at 6 months from the baseline was confirmed to be within the target blood pressure range according to the 2022 hypertension treatment guidelines for essential hypertension patients who received the study drug.

Secondary purpose:

1. Evaluate the efficacy by comparing the change in blood pressure for each drug pattern (monotherapy or combination therapy) at 6 months after administration of the drug to be studied in patients with essential hypertension.
2. Evaluate the safety by checking the incidence (%) of adverse events after administration of the drug to be studied in patients with essential hypertension.
3. Evaluate the safety by checking the peripheral edema incidence rate (%) after administration of the drug to be studied in patients with essential hypertension.
4. Evaluate the safety by checking the headache incidence rate (%) after administration of the drug to be studied in patients with essential hypertension.

ELIGIBILITY:
Inclusion Criteria:

1. Adults over 19 years of age
2. A person who was diagnosed with essential hypertension at the time of participation in the study or was previously diagnosed with essential hypertension and is taking antihypertensive drugs for treatment (Essential hypertension: Systolic blood pressure greater than 140mmHg or diastolic blood pressure greater than 90mmHg)
3. A person whose prescription for the study drug under study was confirmed at the time of participation in the study
4. A person who voluntarily decided to participate in this observational study and gave written consent to the consent form

Exclusion Criteria:

1. Patients who are contraindicated in administration of study drug according to the permission

   * Patients with a history of hypersensitivity to the study drug or its components or other dihydropyridine-based drugs
   * Women who are pregnant or may be pregnant, and women who are lactating
   * Patients with shock (including cardiogenic shock), severe aortic valve stenosis, unstable angina, within 1 month after myocardial infarction, severe hypotension, severe liver dysfunction
2. Patients who are inappropriate to participate in the study in the judgement of the investigator

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with essential hypertension who received Lodien Tab.
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2023-02-22 (Actual); Primary Completion 2025-04-22 (Estimated); Study Completion 2025-07-25 (Estimated)

PRIMARY OUTCOMES:
The ratio(%) of patients whose blood pressure measured at 6 months from the baseline was confirmed to be within the target blood pressure range according to the 2022 hypertension treatment guidelines | after 6 months of prescription for S-Amlodipine compared to baseline
  The ratio(%) of patients whose blood pressure measured at 6 months from the baseline was confirmed to be within the target blood pressure range according to the 2022 hypertension treatment guidelines for essential hypertension patients who received the study drug

CONTACTS AND LOCATIONS:
Locations (1):
- Bundang Seoul University Hospital, Seongnam-si, Gyeonggi-do, South Korea